CLINICAL TRIAL: NCT04529031
Title: Clinical and Biomolecular Characteristics of Reminder-Focused Positive-Psychiatry in Adolescent With Posttraumatic Stress Disorder
Brief Title: Biomolecular Characteristics of Reminder-Focused Positive-Psychiatry
Acronym: RFPP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Naser Ahmadi, MD, PhD, Assistant Professor of Psychiatry, University of California, Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB#20-000444
Record Dates: First submitted 2020-08-20; First posted 2020-08-27 (Actual); Last update posted 2025-01-30 (Actual); Status verified 2025-01

CONDITIONS: Posttraumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RFPP group intervention (Active Comparator): The focus of RFPP is on enhancing contextual discrimination and emotional regulation, and promoting the use of adaptive coping strategies in response to trauma reminders, including recognizing reminders, shifting attention from intrusive memories during exposure to reminders to a focus on positive feelings, thoughts, goals, and choices.
  Interventions: Behavioral: Reminder Focused Positive Psychiatry
- attentional control condition (group process) (Sham Comparator): Subjects will receive progressive muscle relaxation and other relaxation techniques as well as education about PTSD and supportive psychotherapy. Parents will receive 4 sessions of relaxation techniques.
  Interventions: Behavioral: attentional control condition (group process)

INTERVENTIONS:
Behavioral: Reminder Focused Positive Psychiatry — The focus of RFPP is on enhancing contextual discrimination and emotional regulation, and promoting the use of adaptive coping strategies in response to trauma reminders, including recognizing reminders, shifting attention from intrusive memories during exposure to reminders to a focus on positive feelings, thoughts, goals, and choices
  Other Names: Subjects will receive progressive muscle relaxation and other relaxation techniques as well as education about PTSD and supportive psychotherapy
  Arms: RFPP group intervention
Behavioral: attentional control condition (group process) — This group process will undergo telehealth relaxation therapy twice a week for 6-week. Subjects will receive progressive muscle relaxation and other relaxation techniques as well as education about PTSD and supportive psychotherapy
  Other Names: focused relaxation intervention
  Arms: attentional control condition (group process)

SUMMARY:
Objective: Posttraumatic stress disorder (PTSD) is a prevalent neuropsychiatric disorder in children and is associated with increased neurovascular inflammation, suicidality, adulthood mental health disorder, and major adverse events. Reminder focused positive psychiatry (RFPP) has been shown as well tolerated feasible trauma focused intervention that is associated with improved core PTSD symptoms, decreased severity of reactivity to PTSD trauma reminders, and increased vascular function. This study evaluates the clinical and biomolecular characteristics of RFPP in adolescents with PTSD.

Research Design/Overall Impact: After obtaining parents' informed consent and adolescent's assent, 60 adolescents aged 11-15 years old with PTSD, and free of known medical and other major psychiatric disorders will be recruited from the pool of eligible adolescents at Olive View UCLA Pediatrics Clinics (>3000 adolescents with PTSD). Eligible adolescents will be randomized to 1) RFPP group intervention, or 2) an attentional control condition (group process). Thirty subjects in each group will receive twice weekly telehealth intervention of either RFPP or group process, for 6 weeks, and undergo 4 blinded neuropsychiatric assessments at baseline, 3, 6, and 24 weeks. Parents will receive weekly interventions of either positive psychoeducation or group process, for 6 weeks and undergo baseline, 3, 6- and 24-weeks neuropsychiatric assessment. Vascular function, inflammatory biomarkers including CRP, homocysteine, and stress involved gene expression biomarkers (i.e. changes in gene expression of FKBP5, DDX6, B2M, LAIR1, RTN4, NUB1, and a multi-gene Conserved Transcriptional Response to Adversity score (CTRA) will be measured at baseline and 6-week. The primary and secondary endpoints are a) changes in PTSD core and reactivity to trauma reminder severity score in response to RFPP intervention, b) changes in wellbeing, biopsychosocial trait, vascular function, neuroinflammation and gene expression biomarkers in response to RFPP, and c) changes in parents' wellbeing and biopsychosocial trait as well as child-parent interactions.

ELIGIBILITY:
Inclusion Criteria:

* Boy/Girl with documented PTSD,
* aged 11- 15 years old,
* able to read/write in English

Exclusion Criteria:

* presence of intellectual disabilities,
* presence of psychotic or self-injurious behavior,
* presence of seizure disorder,
* presence of language disorder,
* presence of eye disorders,
* presence of other neurodevelopmental disorders,
* presence of diagnosis of substance use disorder.

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-12-28 (Estimated); Study Completion 2026-12-28 (Estimated)

PRIMARY OUTCOMES:
To examine the impact of RFPP intervention on core PTSD symptoms | 24 months
  There will be a change in core PTSD symptoms (% ranged from 0-100) after 6-week RFPP intervention, compared to control group

SECONDARY OUTCOMES:
To assess the impact of RFPP on well-being of adolescents with PTSD and their parents | 24 months
  There will be a change in well-being (% ranged from 0-100), posttraumatic growth (% ranged from 0-100), and parent-child interactions (% ranged from 0-100) in adolescents with PTSD who received RFPP, compared to control group
To examine the impact of RFPP on biologic biomarkers, compared to control group | 24 months
  There will be a change in vascular function ((% ranged from 0-100), stress involved gene expression (% ranged from 0-100), C reactive protein (CRP)(% ranged from 0-100) and homocysteine (% ranged from 0-100) in response to RFPP in adolescents with PTSD

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No